CLINICAL TRIAL: NCT04017208
Title: A Phase 1 Single Ascending Intravenous Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ASP2713 in Healthy Subjects
Brief Title: A Study to Assess ASP2713 in Healthy Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: A business decision was made to not initiate this study.
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2713-CL-0101
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2019-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASP2713 (Experimental): Participants will receive a single dose of ASP2713. Up to 8 dose levels will be administered in the study.
  Interventions: Drug: ASP2713
- Placebo (Placebo Comparator): Participants will receive a single dose of placebo.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ASP2713 — Administered intravenously
  Arms: ASP2713
Drug: placebo — Administered intravenously
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety and tolerability of ASP2713 in healthy participants. The study will also evaluate the pharmacokinetics and pharmacodynamics of ASP2713.

DETAILED DESCRIPTION:
This study will consist of a screening period, a single residential period of 10 days/9 nights and a safety follow up period. Subjects will be randomized to either ASP2713 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index range of 18.5 to 32.0 kg/m^2, inclusive and weighs at least 50 kg at screening.
* Subject has absolute total B cell counts above the lower limit of normal (LLN) reference range measured by flow cytometry at both screening visits 1 and 2. When B cell count reduction (> 50% reduction from the lowest screening baseline value lasting > 6 days postdose in > 4 subjects within a cohort) is observed in a previously enrolled cohort, the subsequent cohorts will enroll only subjects with screening B cell counts above the median of the reference range, as defined by the laboratory.
* Female subject is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance starting at screening and for at least 90 days after study drug administration
* Female subject must agree not to breastfeed 90 days prior to screening and throughout the study period and for 90 days after study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period and for 90 days after study drug administration.
* Male subject with a female partner(s) of childbearing potential must agree to use contraception during the treatment period and for at least 90 days after study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period and for 90 days after study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner(s) is(are) breastfeeding throughout the study period and for 90 days after study drug administration.
* Subject agrees not to participate in another interventional study while participating in the present study, defined as signing of the informed consent form until completion of the last study visit.

Exclusion Criteria:

* Female subject who has been pregnant within 6 months prior to screening or breastfeeding within 3 months prior to screening.
* Subject has known or suspected hypersensitivity to ASP2713 or any components of the formulation used.
* Subject has had previous exposure with ASP2713.
* Subject has any of the liver function tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase and total bilirubin [TBL]) above the upper limit of normal (ULN) at screening visit 1 or on day -2. In such a case, the assessment may be repeated once.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, asymptomatic seasonal allergies) prior to study drug administration.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to day -1.
* Subject has any clinically significant abnormality on physical examination, electrocardiogram (ECG) and clinical laboratory tests at screening visit 1 or day -2.
* Subject has a mean pulse < 45 or > 90 bpm; mean systolic blood pressure > 140 mmHg; mean diastolic blood pressure > 90 mmHg (measurements taken in triplicate after subject has been resting in the supine position for 5 minutes; pulse will be measured automatically) at screening visit 1 or on day -2. If the mean blood pressure exceeds the limits above, 1 additional triplicate measurement can be taken.
* Subject has a mean corrected QT interval using Fridericia's formula (QTcF) of > 430 msec (for male subjects) and > 450 msec (for female subjects) at screening visit 1 or on day -2. If the mean QTcF exceeds the limits above, 1 additional triplicate electrocardiogram (ECG) can be taken.
* Subject has used any prescribed or nonprescribed drugs (including vitamins, natural and herbal remedies, e.g., St John's Wort) in 2 weeks prior to study drug administration, except for occasional use of acetaminophen (up to 2 g per day), hormonal contraceptives or hormone replacement therapy.
* Subject has smoked or has used tobacco-containing products and nicotine or nicotine-containing products within 6 months prior to screening.
* Subject has a history of consuming more than 14 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within the past 2 years prior to screening (note: 1 unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits/hard liquor) or the subject tests positive for alcohol or drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates) at screening or on day -2.
* Subjects has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine and opiates) within 3 months prior to day -2.
* Subject has had significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to day -1.
* Subject has a positive serology test for hepatitis B surface antigen, hepatitis A virus antibodies (immunoglobulin M), hepatitis C virus antibodies, hepatitis B core antibodies or antibodies to human immunodeficiency virus type 1 and/or type 2 at screening.
* Subject has a positive tuberculosis blood test, Quantiferon Gold® or T-SPOT® test at screening.
* Subject has received any vaccine within 60 days prior to study drug administration.
* Subject has received any systemic immunosuppressant agent within 2 months prior to study drug administration.
* Subject has previously received any antibody or therapeutic biologic product 6 months prior to study drug administration.
* Subject has received any systemic steroid within 2 months prior to study drug administration.
* Subject has participated in any clinical study or has been treated with any investigational drugs within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Subject has an absolute lymphocyte count below LLN at screening.
* Subject has any condition which makes the subject unsuitable for study participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to 90 days
  An AE is any untoward medical occurrence in a subject administered a study drug, and which does not necessarily have to have a causal relationship with this treatment. Adverse event (AE) is considered "serious" if the investigator or sponsor view any of the following outcomes: Death, life-threatening, persistent or significant disability/incapacity, congenital anomaly or birth defect, hospitalization, or medically important event. Treatment Emergent Adverse Event (TEAE) is defined as any AE which starts, or worsens, after the first dose of study drug through 30 days after the last dose of study drug.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) [related to treatment] | Up to 90 days
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and /or adverse events (AEs) [related to treatment] | Up to 90 days
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiogram (ECG) abnormalities and/or adverse events (AEs) | Up to 90 days
  Number of participants with potentially clinically significant ECG values.
Number of participants who develop anti-drug antibodies (ADA) to ASP2713 | Up to 90 days
  Number of participants with presence of ADA will be assessed.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ASP2713 in serum: Area under the concentration-time curve (AUC) from the time of dosing extrapolated to time infinity (AUCinf) | Up to 90 days
  AUCinf will be recorded from the pharmacokinetic (PK) serum samples collected.
PK of ASP2713 in serum: AUC from the time of dosing to the last measurable concentration (AUClast) | Up to 90 days
  AUClast will be recorded from the PK serum samples collected.
PK of ASP2713 in serum: AUC extrapolated from time to infinity as a percentage of total area under the concentration-time curve (AUCinf(%extrap)) | Up to 90 days
  AUCinf (%extrap) will be recorded from the PK serum samples collected.
PK of ASP2713 in serum: Maximum concentration (Cmax) | Up to 90 days
  Cmax will be recorded from the PK serum samples collected.
PK of ASP2713 in serum: Clearance (CL) | Up to 90 days
  CL will be recorded from PK serum samples collected.
PK of ASP2713 in serum: Time point prior to the time point corresponding to the first measurable (non-zero) concentration (tlag) | Up to 90 days
  tlag will be recorded from PK serum samples collected.
PK of ASP2713 in serum: Time of the maximum concentration (tmax) | Up to 90 days
  Tmax will be recorded from the PK serum samples collected.
PK of ASP2713 in serum: Terminal elimination half-life (t1/2) | Up to 90 days
  t1/2 will be recorded from PK serum samples collected.
PK of ASP2713 in serum: Apparent volume of distribution during the terminal phase (Vz) | Up to 90 days
  Vz will be recorded from PK serum samples collected.
Pharmacodynamics assessed by ASP2713 receptor occupancy | Up to 90 days
  Blood samples will be collected to measure how much ASP2713 binds to the target on the cell surface.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.